CLINICAL TRIAL: NCT06190782
Title: Phase III Randomized-controlled Study of PD-1 Inhibitor Combined With Local Therapy in Patients With Oligometastatic Esophageal Squamous Cell Carcinoma
Brief Title: Local Therapy for Oligometastatic ESCC Patients Treated With PD-1 Inhibitor
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Kuai Le Zhao, MD, professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESO-Shanghai20
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Esophageal Squamous Cell Carcinoma; Oligometastatic Disease; Radiotherapy
Keywords: esophageal squamous cell carcinom; Oligometastatic; Radiotherapy; pd-1 inhibitor
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD-1 inhibitor+/- chemotherapy combined with local therapy (Experimental): Patients randomized to this arm will receive local treatment combined with systemic treatment (immunotherapy or chemo-immunotherapy)
  Interventions: Combination Product: PD-1 inhibitor+/- chemotherapy combined with local therapy
- PD-1 inhibitor +/- chemotherapy alone (Active Comparator): Patients randomized to this arm will receive only systemic treatment (immunotherapy or chemo-immunotherapy)
  Interventions: Drug: systemic therapy alone

INTERVENTIONS:
Combination Product: PD-1 inhibitor+/- chemotherapy combined with local therapy — 1. PD-1 inhibitor +/- Chemotherapy PD-1 inhibitor: all FDA approved PD-1 inhibitor producter is suitable
     First line:
     i. TP: paclitaxel 135-175mg/m2,d1+ DDP25mg/m2, d1-3 or 75mg/m2,d1;q21d (albumin-bound paclitaxel or paclitaxel liposomes as alternative of paclitaxel permitted as alternative) or ii. PF: DDP Second line (other platinum-based agents permitted as alternative such as carboplatin, nedaplatin, oxaliplatin, lobaplatin, etc.) i. Docetaxel or ii. Irinotecan or iii. Paclitaxel (albumin-bound paclitaxel or paclitaxel liposomes as alternative of paclitaxel permitted as alternatives)
  2. Local therapy i. Radiotherapy GTV=all suspected lesions. SBRT: for lung, liver, adrenal gland, celiac lymphnode metatstases 48Gy/6fx; for spine metastatic disease 30Gy/10Fx; for brain metastases 24Gy/30fx; IMRT: for bone metastatic disease 30Gy/10fx; for esophageal lesion or lesion unsuitable of SBRT 50.4Gy/28fx; ii. Surgery iii. Radiofrequency/microwave ablation
  Arms: PD-1 inhibitor+/- chemotherapy combined with local therapy
Drug: systemic therapy alone — 1.PD-1 inhibitor +/- Chemotherapy PD-1 inhibitor: all FDA approved PD-1 inhibitor producter is suitable
  First line:
  i. TP: paclitaxel 135-175mg/m2,d1+ DDP25mg/m2, d1-3 or 75mg/m2,d1;q21d (albumin-bound paclitaxel or paclitaxel liposomes as alternative of paclitaxel permitted as alternative) or ii. PF: DDP Second line (other platinum-based agents permitted as alternative such as carboplatin, nedaplatin, oxaliplatin, lobaplatin, etc.) i. Docetaxel or ii. Irinotecan or iii. Paclitaxel (albumin-bound paclitaxel or paclitaxel liposomes as alternative of paclitaxel permitted as alternatives)
  Other Names: the systemic therapy only
  Arms: PD-1 inhibitor +/- chemotherapy alone

SUMMARY:
Patients with oligometastatic squamous cell carcinoma were enrolled and randomly assigned to receive either PD-1 inhibitor +/- chemotherapy combined with local therapy or PD-1 inhibitor +/- chemotherapy alone.

The primary end point was progression-free survival (PFS). The secondary end points included overall survival, side effects and local control.

DETAILED DESCRIPTION:
Patients with oligometastatic squamous cell carcinoma were enrolled and 2:1 randomly assigned to receive either PD-1 inhibitor +/- chemotherapy combined with local therapy (radiotherapy, surgery, radiofrequency/microwave ablation, etc.) or PD-1 inhibitor +/- chemotherapy alone. Different local therapy techniques are allowed to be used on different lesions in the same patient.All suspected malignant lesion should be included in local treatment planning in principle.

The primary end point was progression-free survival (PFS). The second end points included overall survival, side effects and local control.

ELIGIBILITY:
Inclusion Criteria:

* 1. ≥18 years old; 2. ECOG 0-1; 3. Esophageal squamous cell carcinoma 4. ASTRO/ESTRO defined genuine oligometastatic disease and consistent with: i. ≤4 distant metastases, ii. ≤3 metastatic lesions within a single organ, iii. maximum diameter of each metastatic lesion ≤5cm; 5. ≥1 pathologically diagnosed metastases

Exclusion Criteria:

* 1. History of disseminated metastases or ASTRO/ESTRO defined induced oligometastatic disease 2.Esophageal perforation/hemorrhage 3.Progression disease after PD-1 inhibitor treatment 4.In-field recurrence 5.Intolerance to chemotherapy or immunotherapy 6.lung V20>25%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Estimated)
Dates: Start 2022-09-27 (Actual); Primary Completion 2025-09-27 (Estimated); Study Completion 2027-09-27 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival difference of PD-1 inhibitor+radiotherapy and PD-1 inhibitor alone | 3-year
  The time between the start of the study treatment(day 1) and progression disease(PD)

SECONDARY OUTCOMES:
overall survival difference of PD-1 inhibitor+radiotherapy and PD-1 inhibitor alone | 3-year
  The time between the start of the study treatment(day 1) and death from an cause or last follow-up for patients alive at the end of the study
treatment related side effect | acute side effects within 3 months, late side effects for 3 months later
  Record the treatment related side effects including acute and late side effects
local control rate | 1-year, 3-year
  the portion of patients who do not develop progression disease or exacerbation of clinical symptoms despite stable disease

CONTACTS AND LOCATIONS:
Overall Officials: Kuaile Zhao, MD, Study Director — Fudan University
Locations (1):
- Fudan University Shanghai cancer center, Shanghai, China

REFERENCES:
- [Derived] Mao G, Xin Z, Fan Q, Zhu H, Ye J, Zhou L, He Y, Xu B, Chen C, Li Z, Gu X, Li X, Wang X, Guo J, Xu Z, Wan P, Zhang Y, Zhang F, Huang C, Yi Q, Huang J, Liang S, Chen J, Lin Y, Fang Q, Chen Y, Ai D, Zhu H, Hao S, Liu Q, Zhao K. ESO-Shanghai 20: phase III clinical trial of anti-PD-1 therapy with local intervention for oligometastatic ESCC. Future Oncol. 2025 Aug;21(20):2575-2584. doi: 10.1080/14796694.2025.2534770. Epub 2025 Jul 30. PMID 40734507